CLINICAL TRIAL: NCT01874782
Title: Transcranial Electrical Stimulation for Management of Orthostatic Instability in Acute Cervical Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Patricia Mills, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12-03534
Record Dates: First submitted 2013-02-12; First posted 2013-06-11 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Orthostatic Hypotension; Postural Hypotension
Keywords: spinal cord injury; cardiovascular; orthostatic hypotension; transcranial electrical stimulation; electrotherapy
MeSH Terms: conditions — Hypotension, Orthostatic; Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial electrical stimulation (Experimental): Subject will be determined as autonomically complete or incomplete injury with measuring of the sympathetic skin responses (SSR+), an established protocol for measuring integrity of sympathetic spinal pathways, versus complete autonomic injury (SSR-).
  Interventions: Device: transcranial electrical stimulation

INTERVENTIONS:
Device: transcranial electrical stimulation — TES: medical device TRANSAIR: electrodes placed on the forehead and over the mastoid processes using Velcro straps. Treatment protocol: six 30-minute sessions over a two-week period and stimulation variables (bipolar current; 1.0-3.0 milliamp (mA) amplitude, 3.5 ms duration and 77.5 Hz frequency).
  Other Names: TRANSAIR (TES Center, St Petersburg, Russia)

SUMMARY:
Individuals with acute cervical spinal cord injury (SCI) can suffer from an excessive and prolonged fall in blood pressure when assuming an upright position, such as transitioning from lying to sitting or standing, a condition also known as orthostatic hypotension (OH). Due to a decrease in cerebral oxygenation, affected individuals can develop debilitating symptoms including lightheadedness, blurred vision, fatigue and even loss of consciousness. Recent evidence suggests that OH has a negative impact on cognition in individuals with SCI. Clinical observations suggest that OH can lead to neurological deterioration in individuals who may otherwise have a stable SCI. The presence of symptomatic OH prevented participation in 43% of physical therapy treatment sessions in a study of individuals with acute SCI despite the use of current treatment options. OH is known to adversely affect health, delay rehabilitation and prolong hospitalization in the acute phase of management of individuals who display it. Our team found OH was present in 41 of 55 (75%) patients with acute cervical SCI at our center in 2004.

We plan to research the efficacy of a low-cost, non-invasive device known as transcranial electrical stimulation (TES) to manage OH in individuals with acute cervical SCI. Previous studies have shown that this device is safe to use in individuals with SCI, and has improved blood pressure control in non-SCI individuals.

We hypothesize that in individuals with acute cervical SCI and OH, TES intervention will elicit an attenuation of the drop in systolic BP (SBP)in response to orthostatic stress. TES-induced differences will be most pronounced in those individuals with sparing of spinal autonomic pathways

ELIGIBILITY:
Inclusion Criteria:

* medically stable individuals with acute traumatic cervical SCI with OH;
* age 18-65 years;
* able to give informed consent.

OH will be defined as per the American Academy of Neurology Consensus as a decrease in systolic BP ≥ 20 mmHg, or diastolic BP ≥ 10 mmHg when assuming an upright position on the sit-up test, whether or not symptoms occur.

Exclusion Criteria:

* individuals with: any clinically important or unstable medical or psychiatric disorders;
* history of seizures;
* neuropsychiatric comorbidity;
* acute conditions that could exacerbate cardiovascular control, ie: untreated urinary tract or chest infections, open wounds, etc;
* alterations in head computed tomography or head MRI;
* any cognitive dysfunction or language barrier that would prevent subjects from following English instructions.
* Use of short acting medications for OH (ie: midodrine) will not be a contra-indication as they will be withheld prior to testing, however having continuous administration of vasopressors will be an exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in orthostatic decrease in BP in response to six sessions of TES, determined via the established bedside sit-up test | The change in BP will be measured between time points: 1. immediately before first TES session and 2. immediately after last TES session.
  In brief, the subject will receive six sessions of thirty minutes duration of transcranial electrical stimulation. Immediately after the last session, the subject will be monitored via finger BP cuff in the supine position for 10 minutes resting BP. Next the subject will be transferred to the sit-up position with continuous BP recording. The decline in BP at three minutes (orthostatic decrease) following assumption of the sit-up posture will be documented.

SECONDARY OUTCOMES:
Long term change in BP. | Change in BP between timepoints 1. immediately before first TES session and 2. 3 weeks after last TES session.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia B Mills, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Center - Vancouver Coastal Health Research Institute, Vancouver, British Columbia, Canada